CLINICAL TRIAL: NCT05587907
Title: The Effect of an Exercise Program With Visual Stimuli on Reaction Time, Cognitive Function and Physical Fitness of Children and Adolescent Soccer Players
Brief Title: Reaction Time, Cognitive Function and Physical Fitness of Children and Adolescent Soccer Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Evangelia Kouidi, Professor of Sports Medicine, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 68/2021
Record Dates: First submitted 2022-09-29; First posted 2022-10-20 (Actual); Last update posted 2022-10-20 (Actual); Status verified 2022-10

CONDITIONS: Neuroplasticity
Keywords: Reaction Time; Cognitive Function; Physical Fitness; FITLIGHT Trainer; Visual Field; VR; soccer players
MeSH Terms: interventions — Exercise Test

STUDY DESIGN:
Intervention Model Description: Around half of the participants follow a 6-month exercise program with visual stimuli, 5 times a week and lasting 15 minutes each time, which precedes their regular soccer training program. The other half of the participants will continue their regular soccer training program. After the end of the 6 months, the initial measurements will be repeated in both groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): 18 soccer players follow a 6-month exercise program with visual stimuli, 5 times a week and lasting 15 minutes each time, which precedes their regular soccer training program.
  Interventions: Device: FitLight Trainer
- Group 2 (No Intervention): 20 soccer players follow a regular soccer training program.

INTERVENTIONS:
Device: FitLight Trainer — Evaluation of the reaction time before and after special training program using visual stimuli.
  Other Names: Cognitive Function Scanner Mobile; VR game; Eurofit Physical Fitness Test Battery; ALPHA-Fitness test battery
  Arms: Group 1

SUMMARY:
Investigation of the effect of an exercise program with visual stimuli on reaction time, cognitive function and physical fitness of children and adolescent soccer players.

DETAILED DESCRIPTION:
38 male soccer players aged 10-15 participate in the research voluntarily. A wireless reflex measurement system (FITLIGHT Trainer) is used to measure the response time, a cognitive function test (Cognitive Function Scanner Mobile) is used to assess cognitive function and an interactive virtual reality application (VR game) is used to estimate the visual field. Physical fitness is assessed using ALPHA-Fitness and the Eurofit test batteries. The screening takes place in the soccer field with portable devices. After the initial check, the participants were randomly divided into two equal groups using the program http://www.randomizer.org/.

18 soccer players follow a 6-month exercise program with visual stimuli, 5 times a week and lasting 15 minutes each time, which precedes their regular soccer training program. The special training program includes training using illuminated units / disks. Each unit is activated alternately, and it is deactivated when the trainee passes in front of it or touches it with any part of his body as well as with another object / sports accessory. The remaining players continue their regular soccer training program. After the end of the 6 months, the initial measurements will be repeated in both groups.

ELIGIBILITY:
Inclusion Criteria: male sex, age 10-15 years, soccer experience ≥ 1year

Exclusion Criteria: None

Ages: 10 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 38 (Actual)
Dates: Start 2021-04-21 (Actual); Primary Completion 2021-12-12 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
Reaction time (sec) | 6 months
  VR game, FITLIGHT Trainer
Cognitive function (sec) | 6 months
  Cognitive Function Scanner Mobile

SECONDARY OUTCOMES:
Physical fitness | 6 months
  RFD (kg/sec), Hand grip test (kg), Sit & reach flexibility (cm), Repeated Sprint (sec)

CONTACTS AND LOCATIONS:
Overall Officials: EVANGELIA KOUIDI, PhD, Study Chair — Department of Physical Education and Sports Sciences Aristotle University of Thessaloniki, Greece
Locations (1):
- Laboratory of Sport Medicine, Department of Physical Education and Sports Sciences Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No